CLINICAL TRIAL: NCT01152268
Title: Predictors of Adolescent Sperm Banking: Development of a Profiling and Referral Tool
Brief Title: Sperm Banking Among Adolescents Newly Diagnosed With Cancer: Development of a Profiling and Referral Tool
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: SBANK10; R21HD061296-01A2 (NIH)
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Cancer
Keywords: sperm banking; Adolescent males; Infertility; Adolescents diagnosed with cancer
MeSH Terms: conditions — Neoplasms; Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adolescent Male Participants: Self-report questionnaire data will be collected one time, between Days 1-7 post initiation of cancer therapy(e.g. Days 2-8 of being "on-treatment" for cancer) among eligible participants and their families who enroll on the study. Patients who agree to participate will be asked to complete a battery of paper and pencil questionnaires (which will also be available on-line if preferred) that assess risk/protective factors for sperm banking. When the banking recommendation is "Yes" or "further assessment required," the profiling and referral tool will be given to the family and instructions for completion will be provided. The tool will include a list of key items which will be based on the most influential barriers to banking sperm.

SUMMARY:
Despite the known adverse effects of specific cancer treatments on fertility, only 18-26% of at-risk adolescents and young men cryopreserve sperm prior to cancer treatment in the US: These already less than optimal rates of sperm banking are even lower among adolescents who have increased anxiety at cancer diagnosis, are lower in age and socioeconomic status, of Evangelical religious orientation, or are diagnosed with leukemia/lymphoma: It is not clear why sperm banking is underutilized, particularly in light of the high priority that survivors of childhood cancer place on fertility and the high psychological distress associated with fertility loss. Studies addressing sperm banking among adults with cancer suggest that factors such as poor physician communication and the resulting lack of fertility-risk knowledge by patients contributes to the low frequency of sperm cryopreservation. No well-designed studies have examined risk factors associated with failure to bank sperm among adolescents with cancer, a developmentally distinct population ripe for intervention.

This study plans to enroll 206 adolescent males and 412 parents/guardians.

DETAILED DESCRIPTION:
This study will identify factors predictive of sperm banking/not sperm banking in order to design interventions for increasing fertility preservation among adolescent males newly diagnosed with cancer. Specifically, this study aims to investigate psychological, demographic, developmental, parent/guardian, provider, and medical factors predictive of sperm banking outcomes among at-risk adolescents with cancer. Once these factors have been identified, the study will develop a novel Profiling and Referral Tool. This instrument will ultimately serve as an intervention for both healthcare providers and families through the facilitation of appropriate referrals, and tailored interventions for decreasing barriers to sperm banking. Finally, the feasibility of the Profiling and Referral tool will be evaluated based on provider and family report.

ELIGIBILITY:
Inclusion Criteria:

* Male participants newly diagnosed with cancer.
* Patients must be between 13 years of age (≥ 13 years) and 21 years of age (< 22 years) at time of study enrollment.
* Participant Identified as Tanner stage III or higher.
* Participant identified by his oncologist (or designee) as being at risk for treatment-related infertility.
* Proficiency speaking and reading English or Spanish.
* Cognitive capacity to complete study questionnaires.

Exclusion Criteria:

* Participant previously treated for cancer.
* History of mental retardation or severe cognitive or learning impairment.

Ages: 13 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male Adolescents meeting eligibility criteria will be identified by updated clinic lists that are available across all institutions included in this study. After the review of clinic lists, medical record review, and report from oncologist regarding patient risk for treatment-related infertility, patients meeting study criteria will be recruited consecutively within the time constraints of the available staff. That is, for every opportunity where there is staff available for recruitment, the study team will attempt to enroll the first available patient meeting eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2010-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Investigation of factors predictive of sperm banking outcome | 3 years
  Investigate factors predictive of banking sperm/not banking sperm among at-risk adolescents newly diagnosed with cancer. Psychological, health belief, demographic, developmental, parental/guardian, provider, and medical factors will be tested in models of sperm banking outcome.

SECONDARY OUTCOMES:
Develop and evaluate a Profiling and Referral Tool designed to increase clinical referrals and decrease barriers to sperm banking. | 3 years
  To utilize factors most predictive of sperm banking outcome to develop a brief Profiling and Referral Tool designed to increase sperm banking among teens newly diagnosed with cancer. Implementation of the developed Profiling and Referral Tool will be feasible based on provider and family report.

CONTACTS AND LOCATIONS:
Overall Officials: James Klosky, Ph.D, Principal Investigator — St. Jude Children's Research Hospital
Locations (9):
- United States (8):
  - City of Hope, Duarte, California
  - Mattel Children's Hospital, Los Angeles, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Dana-Farber Cancer Institute/Children's Hospital Boston, Boston, Massachusetts
  - The University of Michigan, Ann Arbor, Michigan
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Klosky JL, Flynn JS, Lehmann V, Russell KM, Wang F, Hardin RN, Eddinger JR, Zhang H, Schenck LA, Schover LR. Parental influences on sperm banking attempts among adolescent males newly diagnosed with cancer. Fertil Steril. 2017 Dec;108(6):1043-1049. doi: 10.1016/j.fertnstert.2017.08.039. PMID 29202957
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols